CLINICAL TRIAL: NCT06350188
Title: Efficacy of Kinesiotape on Treatment of Nonspecific Cardiac Chest Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Huda Badr Abd El Hamed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECM#2024-506
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Nonspecific Cardiac Chest Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): the patient will receive kinsiotape therapy
  Interventions: Other: experimental
- traditional (Active Comparator): the patient will receive traditional therapy
  Interventions: Other: traditional

INTERVENTIONS:
Other: experimental — 15 patients ˃receive kinisio-tape ,2 session / week for 2 weeks. Followed by stretching exercises, they will be assessed pre and immediately post application, after two weeks and follow up after one month
  Arms: experimental
Other: traditional — 15 patients ˃ will receive ischemic pressure release followed by stretching exercises 2 session / week for 2 weeks, will be assessed pre and immediately post application, after two weeks and follow up after one month.
  Arms: traditional

SUMMARY:
purpose of the study To investigate the effect of Kinesio-tape on treatment of nonspecific cardiac chest pain

DETAILED DESCRIPTION:
Nonspecific musculoskeletal chest pain is a major health problem and is a very common and functionally limiting pain complaint. Patients with this problem complain also of significant disability of daily living activities and lost productivity.

The clinical symptom of anterior chest pain generally elicits a long list of diagnoses, when cardiac and pleural conditions are excluded, conditions that affect the musculoskeletal system become important considerations.

The musculoskeletal structures of the thoracic wall and the neck are relatively common sources of chest pain, hypersensitive loci, named myofascial trigger points in the literature, are associated with the Pathophysiology and clinical manifestation of myofascial pain, Rhomboid Muscle trigger point can be a distressing cause of chest pain which can be effectively taken care of by Ischemic compression therapy. Rhomboid muscle trigger points are one of the major causes of nonspecific cardiac chest pain that make the patient seek treatment in different medical health care, but still there is a lake of scientific evidence that supports a particular treatment. Conducting the current study will find an additional solution for this problem.

Kinesio-Taping a technique highly appropriate in patients with soft tissue involvement and plays a major role in the deactivation of trigger points, KT is theorized to have several functions: (1) restoring correct muscle function by supporting weakened muscles, (2) reducing congestion by improving the flow of blood and lymphatic fluid, (3) decreasing pain by stimulating neurological system, (4) correcting misaligned joints by retrieving muscle spasm, and (5) enhancing proprioception through increased stimulation to cutaneous mechanoreceptors

ELIGIBILITY:
Inclusion Criteria:

* 30 subjects from both sexes with nonspecific cardiac chest pain 2- Rhomboid trigger point 3-All subjects range from 7 to 9 on VAS. 4-Age range from 20-35. 5- All subjects will complain from limited shoulder ROM

Exclusion Criteria:

* Acute coronary syndrome/ ischemic heart disease 2-Pleurisy 3-Pulmonary lessons like(COPD) Chronic Obstructive Pulmonary Disease,( COAD) Chronic Obstructive Airway Disease and Bronchiectasis, 4-Costochondritis, ' 5-Teitze syndrome, 6-Chest wall syndrome 7-Rheumatologic conditions, 8-Infections in the chest wall 9-Gastro-intestinal problems and 10-Neoplastic disorders

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-07-22 (Estimated)

PRIMARY OUTCOMES:
PAIN USING VIISUSL ANALOGE SCALE | up to 2 weeks
  cm line with 0 (no pain) and 10 (killing pain). The patient places a mark along the line to detect his chest pain level.

SECONDARY OUTCOMES:
PERSSURE PAIN THRESHOLD | up to 2 weeks
  The pressure algometer is a simple handheld pressure algometer, placed perpendicular to the tissue surface and pressure applied steadily at a constant rate

OTHER OUTCOMES:
SHOULDER RANGE OF MOTION | up to 2 weeks
  digital level inclinometer will used to assess the shoulder ROM .it has an accuracy ± 0.2º for all angles. Measurements were done three times, and an average will be calculated.
shoulder pain and disability | up to 2 weeks
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Huda Badr Abd Elhamed, Cairo, Egypt